CLINICAL TRIAL: NCT05204212
Title: Prospective, Randomized, Controlled, Unblinded, International, Multicentre, Parallel Two Group Trial of Left Atrial Appendage Closure in Patients With Non-valvular Atrial Fibrillation and End-stage
Brief Title: Left Atrial Appendage Closure in Patients With Non-valvular Atrial Fibrillation and End-stage Chronic KIDNEY Disease
Acronym: LAA-KIDNEY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. med. Ingo Eitel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Ingo Eitel, Director, University of Luebeck
Organization: University of Luebeck (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-392
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF): Paroxysmal, Persistent, Permanent
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention (Experimental): Percutaneous closure of the LAA by use of the CE-mark approved LAA exclusion device Amplatzer Cardiac Plug or Amulet followed by dual antiplatelet therapy with aspirin 100mg od and clopidogrel 75 mg od for 3 months. In patients with excessive bleeding risk DAPT duration can be shortened according to the physicians' discretion to a minimum of 6 weeks. Oral anticoagulants are not prescribed in this group.
  Interventions: Other: Left Atrial Appendage closure
- Control intervention (No Intervention): No catheter-based LAA closure. Treatment with best medical care (warfarin or NOAC therapy or other best medical care if (N)OAC therapy is contraindicated).

INTERVENTIONS:
Other: Left Atrial Appendage closure — Percutaneous closure of the LAA
  Arms: Experimental intervention

SUMMARY:
In the proposed event driven trial, LAA closure devices will be compared in a 1:1 randomization to best medical care in AF patients at high risk of stroke and bleeding with ESKD. The trial will allow the use of the CE marked and clinically used LAA device Amplatzer Cardiac Plug and/or Amulet and all approved medical therapies in AF patients with ESKD including vitamin-K antagonists (VKA), NOACs as well as antiplatelet agents or no anticoagulation in excessive bleeding risk.

DETAILED DESCRIPTION:
The purpose of the current study is to evaluate the clinical benefit of percutaneous catheter-based left atrial appendage (LAA) closure in patients with non-valvular atrial fibrillation (NVAF) and end-stage renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to give informed consent
* Documented NVAF (paroxysmal, persistent, or permanent)
* CHA2DS2VASc risk score ≥2
* Chronic kidney disease KDOQI stage 5 (eGFR <15 ml/min/1.73m2) with or without hemodialysis

Exclusion Criteria:

* Absolute contraindication to aspirin and/or clopidogrel
* Comorbidities other than AF requiring chronic (N)OAC therapy e.g. mechanical heart valve prosthesis
* Present LAA thrombus
* Mobile aortic atheroma
* Age ≤18 years
* Patients presenting with pregnancy
* Patients without informed consent
* Participation in another trial
* Expected life expectancy <2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-01-14 (Estimated); Study Completion 2028-01-14 (Estimated)

PRIMARY OUTCOMES:
"Net clinical benefit" | Day 0
  "Net clinical benefit", defined as, time to first stroke (including ischemic or hemorrhagic strokes), systemic embolism, cardiovascular or unexplained death or major bleeding (BARC 3-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Universität zu Lübeck, Lübeck, Schleswig-Holstein, Germany